CLINICAL TRIAL: NCT05687695
Title: Core Muscle Response to Backward Walking in Patients With Non Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Amr Ahmed Mohammed, assistant lecturer of biomechanics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003264
Record Dates: First submitted 2022-12-22; First posted 2023-01-18 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Non-specific Low Back Pain
Keywords: NSLBP

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- backward walking training group (Experimental): six weeks of backward walking training program 3 times per week
  Interventions: Other: backward walking program
- core training group (Active Comparator): six weeks of core training 3 times per week
  Interventions: Other: core training
- control group (No Intervention): patients will not receive any intervention for six weeks

INTERVENTIONS:
Other: backward walking program — six weeks of backward walking program at self selected speed for 30 minutes 3 times per week
  Arms: backward walking training group
Other: core training — six weeks of core training program including curl up, lateral plank on both sides, bird dog exercises done 3 times per week
  Arms: core training group

SUMMARY:
evaluation of core muscles endurance and strength following backward walking training programe

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted at the Isokinetic laboratory, Faculty of Physical Therapy, Cairo University, to investigate the effect of backward walking training on core muscles strength and endurance, pain severity, and disability level in subjects with NSLBP. Sixty females clinically diagnosed with nonspecific low back pain with age range from 18-45 years will participate in the study. They will be randomly assigned into 3 groups according to the received intervention; backward walking group (BWG), core stability group (CSG), and control group (CG). The isokinetic strength of trunk muscles, and hip extensors and abductors will be evaluated in a concentric mode of muscle contraction. McGill's core endurance tests will be used to examine participants' core endurance. The visual analog scale will be used for measuring the pain intensity. The oswestry disability index will be used to assess pain related disability and quality of life in subjects with LBP.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included if they have a history of LBP for more than 6 weeks before the study, or experienced at least 3 episodes of LBP each lasting more than one week, during the year before the study.

Exclusion Criteria:

* Participants will be excluded if they have:

  1. LBP as a result of a specific spinal condition (e.g. spondylolisthesis, or spinal stenosis).
  2. Previous abdominal or spinal surgery.
  3. Serious spinal conditions (e.g., vertebral fracture, tumor or infection).
  4. Severe musculoskeletal deformity (scoliosis or kyphosis).
  5. Inflammatory disorders (e.g. Rheumatoid arthritis).
  6. Radicular symptoms consistent with a disc herniation, or cauda equina syndrome.
  7. Pain and dysfunction in the upper and lower extremity that would interfere with testing.
  8. Current pregnancy.
  9. Marked leg length discrepancy greater than 2 cm.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — there is gender related difference in the incidence of low back pain
Enrollment: 45 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Change in trunk flexors, extensors and hip extensors, abductors muscles strength | measured twice before and after 6 weeks of intervention
  concentric peak torque of trunk flexors and extensors and hip extensors and abductors
Change in core muscles endurance | measured twice before and after 6 weeks of intervention
  core muscles endurance assessed by McGill endurance tests

SECONDARY OUTCOMES:
Change in pain severity assessed by visual analogue scale | measured twice before and after 6 weeks of intervention
  The Visual Analogue Scale will be used for measuring the pain intensity. It consists of a line, 10 cm long, whose ends are labeled as; no pain and very extreme pain. The line is marked for each 1 cm without any label. Patients are simply asked to indicate which point along the line that best represents their pain intensity. The distance from the "no pain" end to the mark made by the patient will be measured as the patient pain intensity score. VAS is a valid and reliable tool for pain measurement
Change in pain related disability and quality of life | measured twice before and after 6 weeks of intervention
  The Oswestry Disability Index 10 criteria will be used to assess the degree of functional impairment includes pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life (if applicable), social life, and travelling. The ODI scores is expressed in percentages and ranges from 0 (minimum disability) to 100 % (maximum disability).
  For each section the total possible score is 5: if the first statement is marked the section score= 0; if the last statement is marked, it= 5. For example, if all 10 sections are completed the score is calculated as follows: 16 (total scored) ÷ 50 (total possible score) x 100 = 32%. If one section is missed or not applicable the score is calculated as follows: 16 (total scored) ÷ 45 (total possible score) x 100 = 35.5%.

CONTACTS AND LOCATIONS:
Overall Officials: Salam M Elhafez, Professor, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No